CLINICAL TRIAL: NCT04401982
Title: Measuring the Effects of Rhopressa on Episcleral and Retinal Blood Flow in Ocular Hypertension and Glaucoma Suspects Using Erythrocyte Mediated Angiography In Vivo
Brief Title: Measuring the Effects of Rhopressa on Episcleral and Retinal Blood Flow in Ocular Hypertension and Glaucoma Suspects
Status: Completed | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Aerie Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Osamah Saeedi, Associate Professor; Glaucoma Division Chief; Director of Clinical Research, University of Maryland, Baltimore
Other Study IDs: HP-00086248
Record Dates: First submitted 2020-05-20; First posted 2020-05-26 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Ocular Hypertension; Suspect Glaucoma
MeSH Terms: conditions — Ocular Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Glaucoma Suspect: Individuals with a diagnosis of glaucoma suspect
  Interventions: Drug: Netarsudil ophthalmic solution 0.02% one drop nightly for 1-2 weeks

INTERVENTIONS:
Drug: Netarsudil ophthalmic solution 0.02% one drop nightly for 1-2 weeks — Netarsudil ophthalmic solution 0.02% one drop nightly for 1-2 weeks will be administered
  Other Names: Rhopressa

SUMMARY:
Rhopressa effectively lowers intra-ocular pressure by improving conventional outflow and decreasing episcleral venous pressure. While this may result in improved episcleral venous flow, current methods to quantify episcleral blood flow in vivo are rudimentary and unable to accurately and precisely determine flow. Proof that Rhopressa effectively increases episcleral venous flow would differentiate it from other medications. Furthermore, this evidence could galvanize interest in the use of Rhopressa after popular Minimally Invasive Glaucoma Surgery (MIGS) procedures. In future studies, MIGS procedures could be used to improve the proximal outflow pathway, and Rhopressa to enhance distal outflow.

Specific Aim:

To determine the effect of Rhopressa on episcleral venous outflow and retinal blood flow in a cohort of treatment-naïve ocular hypertensive and glaucoma suspect patients.

Hypothesis:

Rhopressa increases episcleral venous flow and retinal blood flow from baseline at both 1 hour and 1 week after initiation of therapy.

DETAILED DESCRIPTION:
Need/Relevance:

Rhopressa effectively lowers intra-ocular pressure by improving conventional outflow and decreasing episcleral venous pressure. While this may result in improved episcleral venous flow, current methods to quantify episcleral blood flow in vivo are rudimentary and unable to accurately and precisely determine flow. Proof that Rhopressa effectively increases episcleral venous flow would differentiate it from other medications. Furthermore, this evidence could galvanize interest in the use of Rhopressa after popular Minimally Invasive Glaucoma Surgery (MIGS) procedures. In future studies, MIGS procedures could be used to improve the proximal outflow pathway, and Rhopressa to enhance distal outflow.

Purpose/Aim:

The investigators have developed a technology to accurately and precisely determine episcleral and retinal blood flow in human subjects using ICG labeled erythrocytes via a technique the investigators have coined as Erythrocyte Mediated Angiography (EMA). The investigators propose conducting a pilot study to show the effect of Rhopressa on both improving episcleral blood flow as well as studying its effect on retinal blood flow. With lower intraocular pressure, and correspondingly higher ocular perfusion pressure, Rhopressa may also improve retinal blood flow.

Specific Aim:

To determine the effect of Rhopressa on episcleral venous outflow and retinal blood flow in a cohort of treatment-naïve ocular hypertensive and glaucoma suspect patients.

Hypothesis:

Rhopressa increases episcleral venous flow and retinal blood flow from baseline at both 1 hour and 1 week after initiation of therapy.

To test this hypothesis, the investigators will measure and compare episcleral venous and retinal blood flow at baseline, 1 hour after Rhopressa instillation and 1 week after initiation of Rhopressa.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years of age.
* Patients must have ocular hypertension or be a glaucoma suspect.
* Patients must be treatment naïve without alternative study treatments or previous history of using topical IOP lowering agents.
* Patients must have an IOP of 24-30 mm Hg in the affected eye.
* Patients must have open angles on gonioscopy.
* Patients must be willing and able to comply with the protocol including providing informed consent.
* All patients will have at least one recorded visual field examination within 6 months of enrollment in the study. Visual fields will be assessed using the Hodapp-Andersen-Parish criteria.

Exclusion Criteria:

* Prior intraocular surgery other than uncomplicated cataract surgery.
* Allergy or history of adverse reaction to ICG, shellfish, or Iodine.
* Significant liver disease or uremia.
* Secondary glaucoma including exfoliation glaucoma, pigmentary glaucoma, or history of acute angle closure.
* Greater than 6 diopters of refractive error.
* Moderate or severe visual field deficits as per Hodapp-Anderson-Parish criteria.
* Any condition precluding imaging including reliable visual fields, disc photography, or use of study treatments including media opacity or tilted optic disk.
* Pregnant or nursing patients.

Ages: 18 Years to 88 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from the optometry service and the glaucoma division at the University of Maryland School of Medicine, Department of Ophthalmology. We will establish a cohort of 10 patients comprised of treatment-naïve ocular hypertensive and glaucoma suspect patients with the following eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-02-22 (Actual)

PRIMARY OUTCOMES:
Change in episcleral venous blood flow with Rhopressa | 1 year
  Change in episcleral venous blood flow with Rhopressa as measured using erythrocyte mediated angiography flowmetry.
Change in retinal blood flow in arterioles and venules less than 100 microns with Rhopressa | 1 year
  Change in retinal blood flow in arterioles and venules less than 100 microns with Rhopressa. Retinal blood flow will be measured with erythrocyte mediated angiography flowmetry

CONTACTS AND LOCATIONS:
Overall Officials: Osamah Saeedi, MD, Principal Investigator — University of Maryland, Baltimore
Locations (4):
- United States (4):
  - University of Maryland Medical Center, Baltimore, Maryland
  - University Physicians Inc., Baltimore, Maryland
  - UM Faculty Physicians, Inc. | 5900 Waterloo Crossing, Columbia, Maryland
  - Maryland Eye Consultants and Surgeons, Silver Spring, Maryland